CLINICAL TRIAL: NCT05932563
Title: Study on the Epidemiological Characteristics of Female Different HPV Vaccination in China
Brief Title: Study on the Epidemiological Characteristics of Female HPV Vaccination in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fujian Maternity and Child Health Hospital (Other)
Responsible Party: Principal Investigator, Binhua Dong, Laboratory of Gynecologic Oncology, Fujian Maternity and Child Health Hospital
Other Study IDs: HVAC2301
Record Dates: First submitted 2023-05-26; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Human Papillomavirus Vaccines; Adverse Effect; Epidemiology; China; Woman

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — DNA specimens of exfoliated cervix cells#Peripheral blood sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The HPV vaccine group: For retrospective cohort population: This study will be based on the database with HPV typing results before HPV vaccination, and the epidemiological characteristics such as adverse reaction symptoms after HPV vaccination in this population will be followed up by telephone or face-to-face, and 1 cervical exfoliated cell and 1 peripheral blood tube will be collected within 1-12 months after HPV vaccination.
  For the prospective cohort:
  All subjects will be enrolled at the time of the first dose of HPV vaccine, followed up 30-60 days after the last dose of HPV vaccine and 12 months after the last dose of HPV vaccine. One cervical exfoliated cell was collected at enrollment and two follow-up visits, and one peripheral blood tube was collected at 30-60 days follow-up after the last dose of HPV vaccine.
- Unvaccinated HPV group: Exfoliated cervical cells were collected to test for HPV genotyping, or HPV genotyping results had been available for nearly 1 year prior to enrollment

SUMMARY:
Human papillomavirus (HPV) is currently one of the most common sexually transmitted infections, according to its carcinogenicity is divided into high-risk genotypes and low-risk genotypes, studies have confirmed that carcinogenic HPV type continuous infection leads to higher incidence of condyloma acuminatum and cervical cancer, while increasing the risk of oropharyngeal cancer, vaginal cancer and other related cancers. Human papillomavirus vaccines have been widely used worldwide to prevent cancers of the lower reproductive tract, such as cervical, anal and vulvar cancers. According to the type, it is divided into domestic two-valent (Vantage), imported two-valent (GlaxoSmithKline), four-valent (Merck) and nine-valent (Merck)HPV vaccines. All four vaccines prevent high-risk HPV 16/18 infection, and there are differences between the quadrivalent and nine-valent HPV vaccine prevention genotypes. The protection rate, immunizing target and immunizing procedure of different valence number are slightly different. Studies have shown that after women receive HPV vaccine, the incidence of arm redness, swelling, fever, pain and other adverse reactions is high, often accompanied by menstrual disorders, sleep problems, emotional irritability, fever, dizziness, headache and other adverse reactions. However, the causal relationship between HPV vaccination and symptoms after vaccination at different prices is controversial, and there is little research in this area. Therefore, we intend to design a multicenter, bidirectional cohort study to investigate the relationship between HPV vaccination with different valence numbers and adverse reactions after vaccination in Chinese women, and to further explore the unknown potential factors affecting the protective effect of HPV vaccine.

DETAILED DESCRIPTION:
Based on the database with HPV typing results before HPV vaccination, this study will follow up the population's epidemiological characteristics such as adverse reaction symptoms after HPV vaccination through telephone or face to face, and collect 1 cervical exfoliated cell and 1 peripheral blood tube (5ml) for HPV genotyping detection and HPV neutralizing antibody detection. Meanwhile, participants were recruited in different regions of China for a period of three months. Follow-up was performed at the time of the first dose of HPV vaccine, 1 month after the third dose, and 12 months after the third dose. The corresponding questionnaire was filled in during enrollment and follow-up, and one cervical exfoliated cell was collected at each of the three follow-up visits for HPV genotyping. At the same time, the peripheral blood tubes were collected one month after the third injection to evaluate the effect of HPV vaccine neutralizing antibodies. The multi-center cohort study was conducted to explore the unknown potential factors affecting the protective effect of HPV vaccine, and the relationship between HPV vaccine with different price and adverse reactions after vaccination in Chinese women.

ELIGIBILITY:
Inclusion Criteria:

-

The retrospective cohort must meet the following conditions:

1. HPV typing results before HPV vaccination;
2. Willing to go to the main center of Fujian Provincial Maternal and Child Health Hospital or branch center for free examination.

Prospective cohort population must meet the following conditions:

1. Female, 9-45 years old (sexual life history);
2. In the next two years, I am willing to go to the main center of Fujian Provincial Maternal and Child Health Hospital or sub-centers for free check-ups;
3. Will receive the first dose of HPV vaccine;
4. There is no abnormal psychological or physical condition before HPV vaccination.

Exclusion Criteria:

1. Subjects who have previously received another commercially available HPV vaccine, or participated in a clinical study of HPV vaccine, or participated in a clinical study of another vaccine within the past 6 months;
2. Women who plan to become pregnant within the next two years;
3. Are immune deficient or have been diagnosed with congenital or acquired immunodeficiency, human immunodeficiency virus (HIV) infection, lymphoma, leukemia, systemic lupus erythematosus, SLE, rheumatoid arthritis, juvenile rheumatoid arthritis (JRA), inflammatory bowel disease, or other autoimmune disease, and have received immunosuppressive therapy within the past 6 months;
4. Subjects with a history of epilepsy, psychosis, medically treatable major depression, convulsions or convulsions, or subjects with a family history of psychosis;
5. Subjects with spleen insufficiency, functional spleen insufficiency, and any disease that results in spleen insufficiency or splenectomy;
6. During the follow-up period, they were not willing to return to the main center or sub-center of the Fujian Maternal and Child Health Hospital to collect cervical exuded cells and/or peripheral blood samples, such as 30-60 days or 12 months after the last HPV vaccination.
7. Pregnant or lactating women;
8. Asexual life history;
9. The investigator believes that there are other factors that are not suitable for participants to participate in clinical trials.

Ages: 9 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women 9 to 45 years of age who have a sexual history and are about to receive their first dose of HPV vaccine, or have had HPV genotyping results for nearly 1 year before receiving HPV vaccine.
Sampling Method: Non-Probability Sample
Enrollment: 1700 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Human Papillomavirus (HPV) genotyping tests | Baseline (Before the first dose of HPV vaccination)
  All participants were tested for human oncovirus (HPV) genotyping prior to the first dose of HPV vaccination
Human Papillomavirus (HPV) genotyping tests | one month after the third dose of HPV vaccination
  Prospective cohort subjects underwent Human Papillomavirus (HPV) genotyping tests at one month after the third dose of HPV vaccination
Human Papillomavirus (HPV) genotyping tests | 12-month after the third dose of HPV vaccination
  Prospective cohort subjects underwent Human Papillomavirus (HPV) genotyping tests at 12-month after the third dose of HPV vaccination
HPV vaccine neutralizing antibody detection | one month after the third dose of HPV vaccination
  Prospective cohort subjects were tested for neutralizing antibodies to the HPV vaccine at one month after the third dose of HPV vaccination
Human Papillomavirus (HPV) genotyping tests | 1 to 12 months after the third dose of HPV vaccination
  Participants in the retrospective cohort were tested for human oncovirus (HPV) genotyping 1-12 months after the third dose of HPV vaccination
HPV vaccine neutralizing antibody detection | 1 to 12 months after the third dose of HPV vaccination
  Participants in the retrospective cohort were tested for HPV vaccine neutralizing antibodies 1-12 months after the third dose of HPV vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Pengming Sun, PhD, Study Chair — Fujian Maternity and Child Health Hospital, Affiliated Hospital of Fujian Medical University
Locations (6):
- China (6):
  - Fujian Maternity and Child Health Hospital, Fuzhou, Fujian
  - Fujian Provincial Center for Disease Control and Prevention, Fuzhou, Fujian
  - Fuzhou Shanghai street community health Service center, Fuzhou, Fujian
  - Shenzhen Maternal and Child Health Hospital, Shenzhen, Guangdong
  - Hubei Maternal and Child HealthCare Hospital, Wuhan, Hubei
  - Xiangya Hospital, Central South University, Changsha, Hunan